CLINICAL TRIAL: NCT00030641
Title: Randomized Study of Docetaxel Versus Docetaxel Plus Genasense™ (G3139; Bcl-2 Antisense Oligonucleotide) in Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: Docetaxel With or Without Oblimersen in Treating Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genta Incorporated (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069185; GENTA-GN304; NCI-G01-2046; UCLA-0301058
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-09

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — oblimersen; Docetaxel

INTERVENTIONS:
Biological: oblimersen sodium
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as docetaxel use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of docetaxel by making the tumor cells more sensitive to the drug. It is not yet known if docetaxel is more effective with or without oblimersen in treating non-small cell lung cancer.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of docetaxel with or without oblimersen in treating patients who have relapsed or refractory non-small cell lung cancer that has been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with non-small cell lung cancer treated with docetaxel with or without oblimersen (G3139).
* Compare the proportion of major antitumor responses in patients treated with these regimens.
* Compare the response duration and time to progression in patients treated with these regimens.
* Compare the safety and clinical benefit of these regimens, in terms of changes in performance status and tumor-related symptoms, in these patients.
* Compare the proportion of patients surviving 6 and 12 months after treatment with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to response to prior first-line chemotherapy regimen (progression vs stable disease, partial response, or complete response), ECOG performance status (0-1 vs 2), and prior paclitaxel treatment (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oblimersen (G3139) IV continuously on days 1-7 and docetaxel IV over 1 hour on day 5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease upon completion of 8 courses may receive 8 or more additional courses at physician's discretion.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Upon completion of 8 courses, patients may continue to receive docetaxel off study at physician's discretion.

Patients are followed every 9 weeks for up to 18 months.

PROJECTED ACCRUAL: A total of 280 patients (140 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small lung cancer (NSCLC)

  * Stage IIIB (malignant pleural/pericardial effusion) or IV
  * Relapsed or refractory disease
* Measurable disease that has not been irradiated
* Previously treated with 1, and only 1, cytotoxic chemotherapy regimen in the neoadjuvant, adjuvant, or metastatic setting
* No untreated or symptomatic brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3 (without growth factor support)
* Platelet count at least 100,000/mm^3
* No bleeding or coagulation disorder

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Albumin at least 3.0 g/dL
* PT no greater than 1.5 times ULN OR INR no greater than 1.3
* PTT no greater than 1.5 times ULN
* No chronic hepatitis
* No chronic cirrhosis

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No uncontrolled congestive heart failure

Pulmonary:

* No severe pulmonary disease
* No requirement for oxygen due to pneumonectomy
* No severe pleural effusion secondary to NSCLC

Immunologic:

* HIV negative
* No active infection
* No active autoimmune disease

Other:

* No other concurrent active cancer
* No uncontrolled diabetes mellitus
* No uncontrolled seizure disorder
* No peripheral neuropathy grade 2 or greater
* No active peptic ulcer disease
* No other significant medical disease
* No intellectual, emotional, or physical disability that would preclude study participation
* No neurologic disorders, overt psychosis, mental disability, or evidence of a limited capacity to give informed consent or to comply with study treatment
* No known hypersensitivity to phosphorothioate-containing oligonucleotides
* No history of hypersensitivity to drugs containing the excipient Tween 80 (polysorbate 80)
* Satisfactory venous access for multi-day continuous infusion
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior cytokines or vaccine therapy for NSCLC
* At least 3 weeks since prior immunotherapy or biologic therapy for NSCLC
* No concurrent anticancer biologic therapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for NSCLC
* No prior docetaxel
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent corticosteroids* except for the following conditions:

  * CNS disease
  * Underlying lung disease NOTE: *Dose must be stable or decreasing for at least 4 weeks before study participation

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for NSCLC
* No prior radiotherapy to 25% or more of bone marrow (e.g., whole pelvis)
* No concurrent anticancer radiotherapy

Surgery:

* At least 3 weeks since prior surgery for NSCLC
* No prior organ allograft

Other:

* Recovered from prior therapy
* Prior first-line epidermal growth factor receptors (EGFR) administered with cytotoxic therapy are allowed
* At least 3 weeks since prior investigational drugs
* At least 3 weeks since other prior therapy NSCLC
* No prior anticancer therapy subsequent to the first (and only) prior cytotoxic chemotherapy regimen
* No prior second-line EGFR therapy
* No prior oblimersen (G3139)
* No other concurrent investigational or anticancer therapies
* No concurrent anticoagulation therapy except for warfarin (1 mg/day) for central line prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Braccia, Study Chair — Genta Incorporated
Locations (44):
- United States (35):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Montgomery Cancer Center, Montgomery, Alabama
  - Little Rock Hematology-Oncology Associates, Little Rock, Arkansas
  - East Bay Medical Oncology, Concord, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Medical Oncology Care Associates, Orange, California
  - Pacific Hematology/Oncology, San Francisco, California
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Whittingham Cancer Center, Norwalk, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Georgia Cancer Specialists - Northside Office, Atlanta, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Hematology Oncology Services, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Summit Medical Group, P.A., Summit, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - North General Hospital, New York, New York
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Charleston Cancer Center, Charleston, South Carolina
  - Arlington Cancer Center, Arlington, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Harold Simmons Cancer Center, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Cancer Care, Weatherford, Texas
  - Madigan Army Medical Center, Tacoma, Washington
  - Yakima Regional Cancer Care Center, Yakima, Washington
  - Morgantown Internal Medicine Group, Morgantown, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
- Canada (4):
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - McGill University, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
- Russia (5):
  - Medical Radiological Research Center RAMS, Kaluga Region
  - Russian Academy of Medical Sciences Cancer Research Center, Moscow
  - P.A. Hertzen Research Oncology Institute, Moscow
  - Municipal Oncological Dispensary, Saint Petersburg
  - Petrov Research Institute of Oncology, Saint Petersburg